CLINICAL TRIAL: NCT03391466
Title: A Phase 3, Randomized, Open-Label Study Evaluating the Efficacy of Axicabtagene Ciloleucel Versus Standard of Care Therapy in Subjects With Relapsed/Refractory Diffuse Large B Cell Lymphoma (ZUMA-7)
Brief Title: Study of Effectiveness of Axicabtagene Ciloleucel Compared to Standard of Care Therapy in Patients With Relapsed/Refractory Diffuse Large B Cell Lymphoma
Acronym: ZUMA-7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTE-C19-107; 2017-002261-22 (EudraCT Number)
Record Dates: First submitted 2017-12-21; First posted 2018-01-05 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — axicabtagene ciloleucel; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Axicabtagene Ciloleucel Treatment (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation antigen (CD) 19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0.
  Participants who will achieve a partial response or complete response and subsequently experience disease progression may have an option to receive a second course of conditioning chemotherapy and axicabtagene ciloleucel.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Standard of Care Therapy (Active Comparator): Participants will receive 2 or 3, 21-day cycles of second-line chemotherapy:
  * R-ICE:rituximab 375mg/m^2 before chemotherapy, ifosfamide 5g/m^2 24 hours continuous infusion (CI) on Day 2+mesna, carboplatin area under the curve (AUC)5 Day 2, maximum dose 800mg, etoposide 100mg/m^2/day on Days 1-3;
  * R-ESHAP:rituximab 375mg/m^2 Day 1, etoposide 40mg/m^2/day IV on Days 1-4, methylprednisolone 500mg/day IV on Days 1-4 or 5, cisplatin at 25mg/m^2/day CI Days 1-4, cytarabine 2g/m^2 on Day 5;
  * R-GDP:rituximab 375mg/m^2 Day 1 (or Day 8), gemcitabine 1g/m^2 on Days 1 and 8, dexamethasone 40mg on Days 1-4, cisplatin 75mg/m^2 Day 1 or carboplatin area under the curve (AUC)=5; or
  * R-DHAP:rituximab 375mg/m^2 before chemotherapy, dexamethasone 40mg/day on Days 1-4, high dose cytarabine 2g/m^2 every 12 hours for 2 doses on Day 2 following platinum, cisplatin 100mg/m^2 24 hours CI on Day 1 or oxaliplatin 100mg/m^2.
  Responders will receive high-dose therapy and autologous stem cell transplant.
  Interventions: Drug: Platinum-containing Salvage Chemotherapy

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — Administered intravenously
  Other Names: KTE-C19; axi-cel; Yescarta ®
  Arms: Axicabtagene Ciloleucel Treatment
Drug: Platinum-containing Salvage Chemotherapy — Platinum-containing salvage chemotherapy (Rituximab-ifosfamide, carboplatin, etoposide (R-ICE), Rituximab-dexamethasone, cytarabine, cisplatin,oxaliplatin (R-DHAP), Rituximab-etoposide, methylprednisolone, cisplatin, cytarabine (R-ESHAP), or Rituximab-gemcitabine, dexamethasone, cisplatin/carboplatin (R-GDP) as selected by treating investigator).
  Arms: Standard of Care Therapy
Drug: Cyclophosphamide — Administered intravenously
  Arms: Axicabtagene Ciloleucel Treatment
Drug: Fludarabine — Administered intravenously
  Arms: Axicabtagene Ciloleucel Treatment

SUMMARY:
The goal of this clinical study is to assess whether axicabtagene ciloleucel therapy improves the clinical outcome compared with standard of care second-line therapy in participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
After completing the treatment period, all participants will be followed in the post-treatment follow-up period for up to 5 years. Thereafter, participants who received at least one dose of axicabtagene ciloleucel as protocol therapy will transition to a separate long term follow up (LTFU) study and complete the remainder of the 15-year follow-up assessments within KT-US-982-5968 (NCT05041309).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically proven large B-cell lymphoma (BCL) including the following types defined by World Health Organization (WHO) 2016.

  * Diffuse large B-cell lymphoma (DLBCL) not otherwise specified activated B-cell/ germinal center B-cell (ABC/GCB).
  * High-grade B-cell lymphoma (HGBL) with or without myelocytomatosis oncogene (MYC) and BCL 2 and/or BCL 6 rearrangement.
  * DLBCL arising from follicular lymphoma (FL).
  * T-cell/histiocyte rich large B-cell lymphoma.
  * DLBCL associated with chronic inflammation.
  * Primary cutaneous DLBCL, leg type.
  * Epstein-Barr virus (EBV) + DLBCL.
* Relapsed or refractory disease after first-line chemoimmunotherapy.

  * Refractory disease defined as no complete remission to first-line therapy; individuals who are intolerant to first-line therapy are excluded.

    * Progressive disease (PD) as best response to first-line therapy.
    * Stable disease (SD) as best response after at least 4 cycles of first-line therapy (eg, 4 cycles of R-CHOP).
    * Partial response (PR) as best response after at least 6 cycles and biopsy-proven residual disease or disease progression ≤ 12 months of therapy.
  * Relapsed disease defined as complete remission to first-line therapy followed by biopsy-proven relapse ≤ 12 months of first-line therapy.
* Individuals must have received adequate first-line therapy including at a minimum:

  * Anti-Cluster of Differentiation 20 antigen (CD20) monoclonal antibody unless investigator determines that tumor is CD20 negative, and
  * An anthracycline containing chemotherapy regimen.
* No known history or suspicion of central nervous system involvement by lymphoma.
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1.
* Adequate bone marrow function as evidenced by:

  * Absolute neutrophil count (ANC) ≥ 1000/μl
  * Platelet ≥ 75,000/μl
  * Absolute lymphocyte count ≥ 100/μl
* Adequate renal, hepatic, cardiac, and pulmonary function as evidenced by:

  * Creatinine clearance (Cockcroft Gault) ≥ 60 mL/min.
  * Serum Alanine aminotransferase/Aspartate aminotransferase (ALT/AST) ≤ 2.5 Upper limit of normal (ULN).
  * Total bilirubin ≤ 1.5 mg/dl
  * Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an Echocardiogram (ECHO), and no clinically significant Electrocardiogram (ECG) findings.
  * No clinically significant pleural effusion.
  * Baseline oxygen saturation > 92% on room air.

Key Exclusion Criteria:

* History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (eg cervix, bladder, breast) unless disease free for at least 3 years.
* Received more than one line of therapy for DLBCL.
* History of autologous or allogeneic stem cell transplant.
* Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous antimicrobials for management.
* Known history of infection with human immunodeficiency virus (HIV) or hepatitis B (HBsAg positive) or anti-hepatitis C virus (HCV) positive. If there is a positive history of treated hepatitis B or hepatitis C, the viral load must be undetectable per quantitative polymerase chain reaction (PCR) and/or nucleic acid testing.
* Individuals with detectable cerebrospinal fluid malignant cells or known brain metastases, or with a history of cerebrospinal fluid malignant cells or brain metastases.
* History or presence of non-malignant central nervous system (CNS) disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
* Presence of any indwelling line or drain. Dedicated central venous access catheter such as a Port-a-Cath or Hickman catheter are permitted.
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, New York Heart Association Class II or greater congestive heart failure, or other clinically significant cardiac diseases within 12 months of enrollment.
* History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment.
* History of autoimmune disease, requiring systemic immunosuppression and/or systemic disease modifying agents within the last 2 years.
* History of anti-Cluster of Differentiation 19 (CD19) or chimeric antigen receptor (CAR)-T therapy or history of prior randomization in ZUMA-7.

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2024-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (72):
- United States (30):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA, Santa Monica, California
  - Stanford Cancer Institute, Stanford, California
  - University of Miami Hospital and Clinics/Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinincs, Iowa City, Iowa
  - The University of Kansas Cancer Center, Kansas City, Kansas
  - University of Maryland, Greenbaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Patient Location, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Henry-Joyce Cancer Center, Nashville, Tennessee
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Swedish Cancer Institute, Seattle, Washington
- Peter MacCallum Cancer Center, Melbourne, Victoria, Australia
- Austria (2):
  - Universitatsklinikum Graz, Division of Hematology, Graz
  - Medizinische Universitat Innsbruck, Innere Medizin V - Hamatologie und Onkologie, Innsbruck
- Belgium (2):
  - Cliniques Universiaires Saint-Luc, Brussels
  - UZ Gasthuisberg, Leuven
- Canada (8):
  - Vancouver General Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Uninversity Health Network - Princess Margaret Cancer Center, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
  - QEII Health Sciences Centre, Halifax
  - Centre Integre Universitaire de Sante et Services Sociaux de l'Est-de-l'lle-de-Montreal / Hopital Maisonneuve-Rosemont, Montreal
  - The Ottawa Hospital - General Campus, Ottawa
  - CHU de Quebec-Universite Laval, Hopital de L'Enfante-Jesus, Québec
- France (4):
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - Hopital Saint-Louis, Paris
  - Centre Hospitalier Lyon-Sud - Service d'Hematologie clinique, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
- Germany (5):
  - Universitäts-klinikum Dresden, Dresden
  - Universitatsmedizin Gottingen, Göttingen
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitäts-klinikum Würzburg, Würzburg
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (2):
  - Instituto di Ematologia "L. e A. Seragnoli" - Dipartimento di Medicina Specialistica Diagnostica e Sperimentale, Bologna
  - IRCCS Ospedale San Raffaele di Milano, Milan
- Netherlands (4):
  - Academic Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
- Uppsala Akademiska Sjukhus, Uppsala, Sweden
- Switzerland (2):
  - IOSI, OSpedale Regionale Bellinzona e Valli, Bellinzona
  - University Hospital Zurich, Zurich
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Barts Health NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Swerdlow SH, Campo E, Pileri SA, Harris NL, Stein H, Siebert R, Advani R, Ghielmini M, Salles GA, Zelenetz AD, Jaffe ES. The 2016 revision of the World Health Organization classification of lymphoid neoplasms. Blood. 2016 May 19;127(20):2375-90. doi: 10.1182/blood-2016-01-643569. Epub 2016 Mar 15. PMID 26980727
- [Background] Elsawy M, Chavez JC, Avivi I, Larouche JF, Wannesson L, Cwynarski K, Osman K, Davison K, Rudzki JD, Dahiya S, Dorritie K, Jaglowski S, Radford J, Morschhauser F, Cunningham D, Martin Garcia-Sancho A, Tzachanis D, Ulrickson ML, Karmali R, Kekre N, Thieblemont C, Enblad G, Dreger P, Malladi R, Joshi N, Wang WJ, Solem CT, Snider JT, Cheng P, To C, Kersten MJ. Patient-reported outcomes in ZUMA-7, a phase 3 study of axicabtagene ciloleucel in second-line large B-cell lymphoma. Blood. 2022 Nov 24;140(21):2248-2260. doi: 10.1182/blood.2022015478. PMID 35839452
- [Background] Kersten MJ, Qiao Y, Shah R, Solem C, Snider JT, To C, Cheng P, Spooner C, Perales MA. Quality-Adjusted Time without Symptoms or Toxicity: Analysis of Axicabtagene Ciloleucel versus Standard of Care in Patients with Relapsed/Refractory Large B Cell Lymphoma. Transplant Cell Ther. 2023 May;29(5):335.e1-335.e8. doi: 10.1016/j.jtct.2023.01.008. Epub 2023 Jan 14. PMID 36646322
- [Background] Locke FL, Miklos DB, Jacobson CA, Perales MA, Kersten MJ, Oluwole OO, Ghobadi A, Rapoport AP, McGuirk J, Pagel JM, Munoz J, Farooq U, van Meerten T, Reagan PM, Sureda A, Flinn IW, Vandenberghe P, Song KW, Dickinson M, Minnema MC, Riedell PA, Leslie LA, Chaganti S, Yang Y, Filosto S, Shah J, Schupp M, To C, Cheng P, Gordon LI, Westin JR; All ZUMA-7 Investigators and Contributing Kite Members. Axicabtagene Ciloleucel as Second-Line Therapy for Large B-Cell Lymphoma. N Engl J Med. 2022 Feb 17;386(7):640-654. doi: 10.1056/NEJMoa2116133. Epub 2021 Dec 11. PMID 34891224
- [Background] Westin JR, Locke FL, Dickinson M, Ghobadi A, Elsawy M, van Meerten T, Miklos DB, Ulrickson ML, Perales MA, Farooq U, Wannesson L, Leslie L, Kersten MJ, Jacobson CA, Pagel JM, Wulf G, Johnston P, Rapoport AP, Du L, Vardhanabhuti S, Filosto S, Shah J, Snider JT, Cheng P, To C, Oluwole OO, Sureda A. Safety and Efficacy of Axicabtagene Ciloleucel versus Standard of Care in Patients 65 Years of Age or Older with Relapsed/Refractory Large B-Cell Lymphoma. Clin Cancer Res. 2023 May 15;29(10):1894-1905. doi: 10.1158/1078-0432.CCR-22-3136. PMID 36999993
- [Background] Westin JR, Oluwole OO, Kersten MJ, Miklos DB, Perales MA, Ghobadi A, Rapoport AP, Sureda A, Jacobson CA, Farooq U, van Meerten T, Ulrickson M, Elsawy M, Leslie LA, Chaganti S, Dickinson M, Dorritie K, Reagan PM, McGuirk J, Song KW, Riedell PA, Minnema MC, Yang Y, Vardhanabhuti S, Filosto S, Cheng P, Shahani SA, Schupp M, To C, Locke FL; ZUMA-7 Investigators; Kite Members. Survival with Axicabtagene Ciloleucel in Large B-Cell Lymphoma. N Engl J Med. 2023 Jul 13;389(2):148-157. doi: 10.1056/NEJMoa2301665. Epub 2023 Jun 5. PMID 37272527
- [Background] Filosto S, Vardhanabhuti S, Canales M, Poiré X, Lekakis LJ, de Vos S, et al. Product attributes of axicabtagene ciloleucel (axi-cel) that associate differentially with efficacy and toxicity in second-line large B-cell lymphoma. Cancer Res. 2022;82(12_Supplement):CT004.
- [Background] Ghobadi A, Munoz J, Westin J, Locke FL, Miklos DB, Rapoport AP, et al. Outcomes of Subsequent Anti-Lymphoma Therapies in Patients (Pts) with Large B-Cell Lymphoma (LBCL) Treated with Axicabtagene Ciloleucel (Axi-Cel) or Standard of Care (SOC) in the Second-Line (2L) ZUMA-7 Study. Blood. 2022;140(Supplement 1):1595-1597.
- [Background] Locke FL, Oluwole OO, Kuruvilla J, Thieblemont C, Morschhauser F, Salles G, et al. Association of Metabolic Tumor Volume (MTV) and Clinical Outcomes in Second-Line (2L) Relapsed/Refractory (R/R) Large B-Cell Lymphoma (LBCL) Following Axicabtagene Ciloleucel (Axi-Cel) Versus Standard-of-Care (SOC) Therapy in ZUMA-7. Blood. 2022;140(Supplement 1):638-640.
- [Background] Chartier M, Filosto S, Peyret T, Chiney M, Milletti F, Budka J, Ndi A, Dong J, Vardhanabhuti S, Mao D, Duffull S, Dodds M, Shen R. Investigating the Influence of Covariates on Axicabtagene Ciloleucel (axi-cel) Kinetics in Patients with Non-Hodgkin's Lymphoma. Clin Pharmacokinet. 2024 Sep;63(9):1283-1299. doi: 10.1007/s40262-024-01413-z. Epub 2024 Sep 6. PMID 39240498
- [Background] Filosto S, Vardhanabhuti S, Canales MA, Poire X, Lekakis LJ, de Vos S, Portell CA, Wang Z, To C, Schupp M, Poddar S, Trinh T, Warren CM, Aguilar EG, Budka J, Cheng P, Chou J, Bot A, Shen RR, Westin JR. Product Attributes of CAR T-cell Therapy Differentially Associate with Efficacy and Toxicity in Second-line Large B-cell Lymphoma (ZUMA-7). Blood Cancer Discov. 2024 Jan 8;5(1):21-33. doi: 10.1158/2643-3230.BCD-23-0112. PMID 37983485
- [Background] Ghobadi A, Munoz J, Westin JR, Locke FL, Miklos DB, Rapoport AP, Perales MA, Reagan PM, McGuirk J, Jacobson CA, Kersten MJ, Avivi I, Peng A, Schupp M, To C, Oluwole OO. Outcomes of subsequent antilymphoma therapies after second-line axicabtagene ciloleucel or standard of care in ZUMA-7. Blood Adv. 2024 Jun 11;8(11):2982-2990. doi: 10.1182/bloodadvances.2023011532. PMID 38315832
- [Background] Locke FL, Chou J, Vardhanabhuti S, Perbost R, Dreger P, Hill BT, et al. Association of pretreatment (preTx) tumor characteristics and clinical outcomes following second-line (2L) axicabtagene ciloleucel (axi-cel) versus standard of care (SOC) in patients (pts) with relapsed/refractory (R/R) large B-cell lymphoma (LBCL). J Clin Oncol.2022;40(16_suppl):7565
- [Background] Locke FL, Filosto S, Chou J, Vardhanabhuti S, Perbost R, Dreger P, Hill BT, Lee C, Zinzani PL, Kroger N, Lopez-Guillermo A, Greinix H, Zhang W, Tiwari G, Budka J, Marincola FM, To C, Mattie M, Schupp M, Cheng P, Bot A, Shen R, Bedognetti D, Miao H, Galon J. Impact of tumor microenvironment on efficacy of anti-CD19 CAR T cell therapy or chemotherapy and transplant in large B cell lymphoma. Nat Med. 2024 Feb;30(2):507-518. doi: 10.1038/s41591-023-02754-1. Epub 2024 Jan 17. PMID 38233586
- [Background] Locke FL, Oluwole OO, Kuruvilla J, Thieblemont C, Morschhauser F, Salles G, Rowe SP, Vardhanabhuti S, Winters J, Filosto S, To C, Cheng P, Schupp M, Korn R, Kersten MJ. Axicabtagene ciloleucel vs standard of care in second-line large B-cell lymphoma: outcomes by metabolic tumor volume. Blood. 2024 Jun 13;143(24):2464-2473. doi: 10.1182/blood.2023021620. PMID 38557775
- [Background] Lunning MA, Wang HL, Hu ZH, Locke FL, Siddiqi T, Jacobson CA, Ahmed S, Miklos DB, Lin Y, Hill BT, Ghobadi A, Neelapu SS, Westin J, Dieyi C, Field P, Miao H, Shahani SA, Patel A, Spooner C, Fu C, Muramoto D, Xu H, Pasquini MC. Benefit of axicabtagene ciloleucel versus chemoimmunotherapy in older patients and/or patients with poor ECOG performance status with relapsed or refractory large B-cell lymphoma after 2 or more lines of prior therapy. Am J Hematol. 2024 May;99(5):880-889. doi: 10.1002/ajh.27283. Epub 2024 Mar 19. PMID 38504387
- [Background] Tian Y, Budka J, Locke FL, Westin JR, To C, Tiwari G, Mao D, Bedognetti D, Shen RR, Andrade J, Filosto S. Tumor gene expression signatures associated with outcome in large B-cell lymphoma treated with CD19-directed CAR T-cell therapy (axicabtagene ciloleucel). Front Oncol. 2025 Feb 27;15:1519473. doi: 10.3389/fonc.2025.1519473. eCollection 2025. PMID 40083872
- [Derived] Locke FL, Siddiqi T, Jacobson CA, Ghobadi A, Ahmed S, Miklos DB, Perales MA, Munoz J, Fingrut WB, Pennisi M, Gauthier J, Shadman M, Gowda L, Mirza AS, Abid MB, Hong S, Majhail NS, Kharfan-Dabaja MA, Khurana A, Badar T, Lin Y, Bennani NN, Herr MM, Hu ZH, Wang HL, Baer A, Baro E, Miao H, Spooner C, Xu H, Pasquini MC. Real-world and clinical trial outcomes in large B-cell lymphoma with axicabtagene ciloleucel across race and ethnicity. Blood. 2024 Jun 27;143(26):2722-2734. doi: 10.1182/blood.2023023447. PMID 38635762
- [Derived] The Lancet Haematology. The role of conferences in tackling inequalities. Lancet Haematol. 2022 Feb;9(2):e81. doi: 10.1016/S2352-3026(22)00008-4. No abstract available. PMID 35114155
- [Derived] Del Pozo Martin Y. 2021 ASH annual meeting. Lancet Haematol. 2022 Feb;9(2):e92-e93. doi: 10.1016/S2352-3026(21)00384-7. Epub 2021 Dec 16. No abstract available. PMID 34922648
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Thiruvengadam SK, Hunter B, Varnavski A, Fakhri B, Kaplan L, Ai WZ, Pampaloni M, Huang CY, Martin T 3rd, Damon L, Andreadis CB. Ofatumumab, Etoposide, and Cytarabine Intensive Mobilization Regimen in Patients with High-risk Relapsed/Refractory Diffuse Large B-Cell Lymphoma Undergoing Autologous Stem Cell Transplantation. Clin Lymphoma Myeloma Leuk. 2021 Apr;21(4):246-256.e2. doi: 10.1016/j.clml.2020.11.005. Epub 2020 Nov 11. PMID 33288485
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KTE-C19-107

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Middle East, Europe, and Australia.
Pre-assignment Details: 437 participants were screened.
Groups:
- Axicabtagene Ciloleucel: Participants received cyclophosphamide 500 mg/m^2/day intravenous (IV) infusion and fludarabine 30 mg/m^2/day IV infusion conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation antigen (CD) 19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0.
- Standard of Care Therapy: Participants received 2 or 3, 21-day cycles of second-line chemotherapy regimen:
  R-ICE: rituximab 375mg/m^2 before chemotherapy, ifosfamide 5g/m^2 24 hours continuous infusion (CI) on Day 2 + mesna, carboplatin area under the curve (AUC) 5 Day 2, maximum dose 800mg, etoposide 100mg/m^2/day on Days 1-3; R-ESHAP: rituximab 375mg/m^2 Day 1, etoposide 40mg/m^2/day IV on Days 1-4, methylprednisolone 500mg/day IV on Days 1-4 or 5, cisplatin at 25mg/m^2/day CI Days 1-4, cytarabine 2g/m^2 on Day 5; R-GDP: rituximab 375mg/m^2 Day 1 (or Day 8), gemcitabine 1g/m^2 on Days 1 and 8, dexamethasone 40mg on Days 1-4, cisplatin 75mg/m^2 Day 1 or carboplatin AUC=5; or R-DHAP: rituximab 375mg/m^2 before chemotherapy, dexamethasone 40mg/day on Days 1-4, high dose cytarabine 2g/m^2 every 12 hours for 2 doses on Day 2 following platinum, cisplatin 100mg/m^2 24 hours CI on Day 1 or oxaliplatin 100mg/m^2.
  Participants who responded to second-line chemotherapy got high dose therapy and autologous stem cell transplant.
Period: Overall Study
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Started | 180 | 179
Completed | 2 | 67
Not Completed | 178 | 112
Not completed — Death | 84 | 91
Not completed — Rollover to Long-term Follow-up Study Criteria | 80 | 0
Not completed — Subject Withdrawal of Consent from Further Follow-up | 3 | 13
Not completed — Lost to Follow-up | 9 | 5
Not completed — Reason Not Specified | 2 | 2
Not completed — Investigator Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all randomized participants.
Groups:
- Axicabtagene Ciloleucel: Participants received cyclophosphamide 500 mg/m^2/day IV infusion and fludarabine 30 mg/m^2/day IV infusion conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD 19 CAR transduced autologous T cells/kg on Day 0.
- Standard of Care Therapy: Participants received 2 or 3, 21-day cycles of second-line chemotherapy regimen:
  * R-ICE: rituximab 375mg/m^2 before chemotherapy, ifosfamide 5g/m^2 24 hours CI on Day 2 + mesna, carboplatin AUC 5 Day 2, maximum dose 800mg, etoposide 100mg/m^2/day on Days 1-3;
  * R-ESHAP: rituximab 375mg/m^2 Day 1, etoposide 40mg/m^2/day IV on Days 1-4, methylprednisolone 500mg/day IV on Days 1-4 or 5, cisplatin at 25mg/m^2/day CI Days 1-4, cytarabine 2g/m^2 on Day 5;
  * R-GDP: rituximab 375mg/m^2 Day 1 (or Day 8), gemcitabine 1g/m^2 on Days 1 and 8, dexamethasone 40mg on Days 1-4, cisplatin 75mg/m^2 Day 1 or carboplatin AUC=5; or
  * R-DHAP: rituximab 375mg/m^2 before chemotherapy, dexamethasone 40mg/day on Days 1-4, high dose cytarabine 2g/m^2 every 12 hours for 2 doses on Day 2 following platinum, cisplatin 100mg/m^2 24 hours CI on Day 1 or oxaliplatin 100mg/m^2.
  Participants who responded to second-line chemotherapy got high dose therapy and autologous stem cell transplant.
- Total: Total of all reporting groups
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy | Total
Number analyzed (Participants) | 180 | 179 | 359
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 129 | 121 | 250
  >=65 years | 51 | 58 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (12.0) | 57.4 (12.2) | 57.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 52 | 122
  Male | 110 | 127 | 237
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 167 | 169 | 336
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 12 | 10 | 22
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 11 | 7 | 18
  White | 145 | 152 | 297
  More than one race | 10 | 8 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 130 | 120 | 250
  United Kingdom | 4 | 8 | 12
  Switzerland | 1 | 0 | 1
  Spain | 6 | 9 | 15
  Canada | 10 | 10 | 20
  Belgium | 4 | 3 | 7
  Netherlands | 11 | 14 | 25
  Sweden | 0 | 1 | 1
  Italy | 2 | 1 | 3
  Israel | 4 | 2 | 6
  Australia | 2 | 2 | 4
  France | 4 | 2 | 6
  Germany | 1 | 5 | 6
  Austria | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS) Per Blinded Central Assessment
Description: EFS:Time from randomization to disease progression (PD), best response of stable disease (SD) up to Day 150, start of new anti-lymphoma therapy including stem cell transplant, or death from any cause. PD=Score 4 (uptake moderately > liver) or 5 (uptake markedly > liver and/or new lesions) with increased uptake from baseline; New fluorodeoxyglucose (FDG)-avid foci consistent with lymphoma rather than another etiology or in bone marrow; Individual node/lesion abnormal with longest diameter > 1.5 cm, ≥ 50% increase from nadir; Splenic length increase > 50% of prior increase beyond baseline or ≥ 2 cm increase if no prior splenomegaly; New/recurrent splenomegaly, progression of non-measurable lesions, new lesion, or new/recurrent bone marrow involvement. KM estimates was used for analysis.
Time Frame: From randomization date up to a median follow-up: 24.9 months
Population: Participants in Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Axicabtagene Ciloleucel: Participants received cyclophosphamide 500 mg/m^2/day IV infusion and fludarabine 30 mg/m^2/day IV infusion conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0.
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 180 | 179
months | 8.3 [4.5 to 15.8] | 2.0 [1.6 to 2.8]
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Test type: Superiority — One-sided p-value based on log-rank test stratified by response to first-line therapy and second-line age-adjusted International Prognostic Index (IPI) as data collected on case report forms; p < 0.0001, Log Rank — Stratified (randomization factors) log-rank p-value; Stratified (randomization stratification factors) log-rank test; Hazard Ratio (HR) = 0.398, 95% CI 2-sided [0.308 to 0.514] — Hazard ratio (95% confidence interval (CI)), stratified using randomization stratification factors

2. Secondary Outcome: Objective Response Rate (ORR) Per Blinded Central Assessment
Description: ORR: Percentage of participants with CR (Complete Metabolic Response (CMR);Complete Radiologic Response (CRR)) or PR (partial metabolic response (PMR); partial radiologic response (PRR)).CMR: Positron emission tomography (PET) 5-point scale scores: 1-No uptake above background; 2-Uptake ≤mediastinum; 3-Uptake >mediastinum but ≤liver, with/without residual mass; no new lesions, no FDG-avid disease in bone marrow. CRR: Target nodes/nodal masses regressed ≤1.5 cm in longest diameter, no extralymphatic sites, no non-measured lesions, normal organ size, no new sites, normal bone marrow morphology. PMR: Scores 4 (uptake moderately >liver), 5 (uptake markedly >liver, new lesions) with reduced uptake from baseline and residual mass, no new lesions. Responding at interim/residual disease at end of treatment. PRR: ≥50% decrease in sum of diameters of up to 6 target measurable lesions, no increase in non-measured lesions, spleen length decreased >50% if previously enlarged, no new lesion sites.
Time Frame: From randomization date up to a median follow-up: 24.9 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 180 | 179
percentage of participants | 83 [77.1 to 88.5] | 50 [42.7 to 57.8]
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Test type: Superiority — One-sided p-value based on Cochran-Mantel-Haenszel (CMH) test, one-sided tailed test, stratified by response to first-line therapy and second-line age-adjusted International Prognostic Index (IPI) as data collected on case report forms; p < 0.0001, Cochran-Mantel-Haenszel — Stratified (randomization factor) CMH test p-value; Stratified (randomization factor) CMH test; Difference in ORR = 33.1, 95% CI 2-sided [23.2 to 42.1] — 95% CI for the difference in ORR was from Wilson's score method with continuity correction

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to death from any cause. Kaplan-Meier (KM) estimates were used for analysis.
Time Frame: Up to 74.9 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 180 | 179
months | NA [28.3 to NA] — Median and upper limit of CI were not reached due to insufficient number of events. | 35.1 [18.5 to NA] — Upper limit of CI was not reached due to insufficient number of events.
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Test type: Superiority — One-sided p-value based on log-rank test stratified by response to first-line therapy and second-line age-adjusted IPI as data collected on case report forms; p = 0.027, Log Rank — Stratified log-rank (randomization factor) p-value; Stratified (randomization factor) log-rank test; Hazard Ratio (HR) = 0.730, 95% CI 2-sided [0.530 to 1.007] — Stratified Cox regression models were used to estimate hazard ratio and 2-sided CIs for axicabtagene ciloleucel relative to standard of care therapy. The Breslow method was used to handle the ties for the Cox regression models; The Rho family spending function with parameter (Rho = 6) was used to allocate alpha between the interim and primary OS analysis. Given that fewer than the anticipated 210 events were observed at the data cutoff date for the primary OS analysis (25 January 2023), the efficacy boundary for the primary OS analysis was recalculated using the Rho family spending function based on the actual observed event numbers (177 deaths) resulting in an efficacy boundary at 1-sided significance level of 0.0249

4. Secondary Outcome: Duration of Response (DOR) Per Blinded Central Assessments
Description: DOR was defined only for participants who experience an objective response after axicabtagene ciloleucel infusion and was the time from the first objective response per Lugano classification to disease progression or death from any cause. Objective response was defined in outcome measure 2 and disease progression was defined in outcome measure 1. KM estimates were used for analysis.
Time Frame: From the date of first confirmed objective response (CR or PR) to disease progression or death regardless of cause (Up to 37.8 months)
Population: Participants in the Full Analysis Set with objective response were analyzed. Participants not meeting the criteria by the analysis data cut-off date were censored at their last evaluable disease assessment date prior to the data cut-off date or new lymphoma therapy start date (including stem cell transplant in the axicabtagene ciloleucel arm or retreatment of axicabtagene ciloleucel), whichever was earlier.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 150 | 90
months | 26.9 [13.6 to NA] — Upper limit of CI was not reached due to insufficient number of events. | 8.9 [5.7 to NA] — Upper limit of CI was not reached due to insufficient number of events.
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0695, Log Rank — Stratified (randomization stratification factors) log-rank test; Hazard Ratio (HR) = 0.736, 95% CI 2-sided [0.488 to 1.108] — Stratified Cox regression models were used to estimate hazard ratio and 2-sided 95% CIs for axicabtagene ciloleucel relative to standard of care

5. Secondary Outcome: Modified Event Free Survival (mEFS) Per Blinded Central Assessment
Description: Modified event free survival is defined the same way as EFS, except that a best response of SD up to and including Day 150 assessment post randomization was not considered an event. KM estimates were used for analysis.
Time Frame: From randomization date up to a median follow-up: 24.9 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 180 | 179
months | 10.3 [5.0 to 21.5] | 2.0 [1.6 to 2.8]
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Test type: Superiority; p < 0.0001, Log Rank — One-sided p-value based on log-rank test stratified by response to first-line therapy and second-line age-adjusted IPI as data collected on case report forms; Stratified (randomization stratification factors) log-rank test; Hazard Ratio (HR) = 0.376, 95% CI 2-sided [0.290 to 0.487] — Stratified Cox regression models were used to estimate hazard ratio and 2-sided 95% CIs for axicabtagene ciloleucel relative to standard of care therapy. The Breslow method was used to handle the ties for the Cox regression models

6. Secondary Outcome: EFS Per Investigator Disease Assessments
Description: EFS was defined as the time from randomization to the earliest date of disease progression per the Lugano Classification, best response of stable disease (SD) up to and including Day 150, commencement of new lymphoma therapy, or death from any cause. Disease progression is defined in outcome measure 1.
Time Frame: From randomization date up to a median follow-up: 47.2 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 180 | 179
months | 10.8 [5.0 to 25.5] | 2.3 [1.7 to 3.1]
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Test type: Superiority; Hazard Ratio (HR) = 0.422, 95% CI 2-sided [0.327 to 0.545] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Progression-Free Survival (PFS) Per Investigator Disease Assessments
Description: PFS is defined as the time from the randomization date to the date of disease progression per Lugano classification or death from any cause. Disease progression is defined in outcome measure 1. KM estimates were used for analysis.
Time Frame: From randomization date up to a median follow-up: 47.2 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 180 | 179
months | 14.7 [5.4 to 43.5] | 3.7 [2.9 to 5.3]
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Test type: Superiority; Hazard Ratio (HR) = 0.506, 95% CI 2-sided [0.383 to 0.669] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Modified Event Free Survival (mEFS) Per Investigator Assessment
Description: mEFS is defined the same way as EFS, except that a best response of SD up to and including Day 150 assessment post randomization was not considered an event. KM estimates were used for analysis.
Time Frame: From randomization date up to a median follow-up: 47.2 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 180 | 179
months | 12.6 [5.0 to 29.1] | 2.3 [1.7 to 3.1]
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Test type: Superiority; Hazard Ratio (HR) = 0.412, 95% CI 2-sided [0.318 to 0.532] — [estimate comment as in outcome 5, analysis 1]

9. Secondary Outcome: Change From Baseline in Global Health Status Scores
Description: Global health status was measured using European Organization for Research and Treatment of Cancer (EORTC) Quality Life Questionnaire (QLQ) C-30. This health related quality of life (HRQoL) questionnaire was comprised of 15 questions on functional scales, 13 questions on symptom scales and 2 on global health status scale. Global Health Status used a 7 point Likert-type scale of 1 (Very poor) to 7 (Excellent). All scores were transformed to 0-100. Higher scores for Global Health Status indicated better HRQoL.
Time Frame: Baseline, Days 50, 100, and 150; Months 9, 12, 15, 18, 21 and 24
Population: Participants in Quality of Life (QoL) Analysis Set with data available at given timepoint were analyzed. The QoL Analysis Set was defined as the subset of participants in the Full Analysis Set who have a baseline and Day 150 post-randomization QoL assessment.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 165 | 130
Score on scale
  Score at Baseline | 68.6 (19.9) | 70.1 (23.1)
  Change from Baseline at Study Day 50: number analyzed (Participants) | 163 | 124
  Change from Baseline at Study Day 50 | -7.4 (20.2) | -8.5 (22.7)
  Change from Baseline at Study Day 100: number analyzed (Participants) | 146 | 62
  Change from Baseline at Study Day 100 | 1.3 (19.6) | -15.3 (22.7)
  Change from Baseline at Study Day 150: number analyzed (Participants) | 110 | 56
  Change from Baseline at Study Day 150 | 5.9 (24.9) | -4.2 (23.7)
  Change from Baseline at Study Month 9: number analyzed (Participants) | 88 | 40
  Change from Baseline at Study Month 9 | 8.0 (22.7) | 3.5 (23.7)
  Change from Baseline at Study Month 12: number analyzed (Participants) | 79 | 33
  Change from Baseline at Study Month 12 | 8.6 (24.9) | 9.1 (20.2)
  Change from Baseline at Study Month 15: number analyzed (Participants) | 67 | 26
  Change from Baseline at Study Month 15 | 9.0 (22.3) | 9.9 (18.9)
  Change from Baseline at Study Month 18: number analyzed (Participants) | 71 | 23
  Change from Baseline at Study Month 18 | 10.2 (20.9) | 6.5 (21.3)
  Change from Baseline at Study Month 21: number analyzed (Participants) | 45 | 20
  Change from Baseline at Study Month 21 | 10.0 (21.5) | 15.0 (19.6)
  Change from Baseline at Study Month 24: number analyzed (Participants) | 32 | 12
  Change from Baseline at Study Month 24 | 8.6 (21.0) | 13.2 (17.2)
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Difference in mean change of scores from Baseline at Day 100; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures — False Discovery Rate Methodology; Mixed Model with Repeated Measures = 18.1, 95% CI 2-sided [12.3 to 23.9]
Statistical Analysis 2: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Difference in mean change of scores from Baseline at Day 150; Test type: Superiority; p = 0.0124, Mixed Model with Repeated Measures — False Discovery Rate Methodology; Mixed Model with Repeated Measures = 9.8, 95% CI 2-sided [2.6 to 17.0]
Statistical Analysis 3: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Difference in mean change of scores from Baseline at Month 9; Test type: Superiority; p = 0.2655, Mixed Model with Repeated Measures — False Discovery Rate Methodology; Mixed Model with Repeated Measures = 4.4, 95% CI 2-sided [-3.3 to 12.0]

10. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Physical Functioning Score
Description: The EORTC QLQ-C30 is composed of global health status/QoL scale; five functional domains (physical, role, emotional, cognitive, and social); three symptom domains (fatigue, nausea and vomiting, and pain); and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties).
  The Physical Functioning domain includes 5 questions in which participants were asked to rate their overall health and overall quality of life as it relates to physical functioning during the past week on a scale from 1 (very poor) to 7 (excellent). The 5 scores were transformed to a scale from 0 to 100, where a high score indicated better QoL. A positive change from baseline indicates better QoL.
Time Frame: Baseline, Days 50, 100, 150, Months 9, 12, 15, 18, 21 and 24
Population: Participants in QoL analysis set with data available at given timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 164 | 131
Score on scale
  Score at Baseline | 83.5 (17.7) | 85.3 (18.9)
  Change from Baseline at Study Day 50: number analyzed (Participants) | 162 | 126
  Change from Baseline at Study Day 50 | -12.9 (21.7) | -8.3 (17.5)
  Change from Baseline at Study Day 100: number analyzed (Participants) | 146 | 64
  Change from Baseline at Study Day 100 | -1.8 (17.8) | -15.0 (19.1)
  Change from Baseline at Study Day 150: number analyzed (Participants) | 109 | 56
  Change from Baseline at Study Day 150 | 1.3 (18.9) | -5.2 (21.3)
  Change from Baseline at Study Month 9: number analyzed (Participants) | 88 | 40
  Change from Baseline at Study Month 9 | 4.1 (17.1) | -2.4 (23.5)
  Change from Baseline at Study Month 12: number analyzed (Participants) | 79 | 33
  Change from Baseline at Study Month 12 | 3.4 (20.8) | 0.4 (20.3)
  Change from Baseline at Study Month 15: number analyzed (Participants) | 67 | 26
  Change from Baseline at Study Month 15 | 3.9 (19.3) | 1.6 (16.1)
  Change from Baseline at Study Month 18: number analyzed (Participants) | 71 | 23
  Change from Baseline at Study Month 18 | 5.0 (15.1) | 3.2 (17.9)
  Change from Baseline at Study Month 21: number analyzed (Participants) | 45 | 20
  Change from Baseline at Study Month 21 | 6.0 (16.1) | 4.3 (21.4)
  Change from Baseline at Study Month 24: number analyzed (Participants) | 32 | 12
  Change from Baseline at Study Month 24 | 3.7 (16.5) | 5.6 (8.0)
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Difference in mean change of scores from Baseline at Day 100; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures — False Discovery Rate Methodology; Mixed Model with Repeated Measures = 13.1, 95% CI 2-sided [8.0 to 18.2]
Statistical Analysis 2: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Difference in mean change of scores from Baseline at Day 150; Test type: Superiority; p = 0.1253, Mixed Model with Repeated Measures — False Discovery Rate Methodology; Mixed Model with Repeated Measures = 5.1, 95% CI 2-sided [-0.9 to 11.0]

11. Secondary Outcome: Changes From Baseline in the European Quality of Life Five Dimensions Five Levels Scale Index Score
Description: The Euro-QOL (EQ) Five Dimensions (5D) Five Levels (5L), EQ-5D-5L questionnaire was a generic measure of health status that provided a simple descriptive profile and a single index value. The EQ-5D-5L comprised 2 components: a questionnaire covering 5 dimensions and a tariff of values based upon direct valuations of health stated using a visual analog scale (VAS). The total score for EQ-5D-5L index was presented on a range from 0 to 1 where higher scores indicated better outcome. A positive change from Baseline indicates improvement.
Time Frame: Baseline, Days 50, 100, 150; Months 9, 12, 15, 18, 21 and 24
Population: Participants in QoL analysis set with data available at given timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 165 | 131
Score on scale
  Score at Baseline | 0.803 (0.210) | 0.799 (0.250)
  Change from Baseline at Study Day 50: number analyzed (Participants) | 163 | 123
  Change from Baseline at Study Day 50 | -0.049 (0.205) | -0.003 (0.198)
  Change from Baseline at Study Day 100: number analyzed (Participants) | 146 | 65
  Change from Baseline at Study Day 100 | 0.012 (0.191) | -0.068 (0.246)
  Change from Baseline at Study Day 150: number analyzed (Participants) | 109 | 56
  Change from Baseline at Study Day 150 | 0.050 (0.212) | 0.014 (0.208)
  Change from Baseline at Study Month 9: number analyzed (Participants) | 88 | 39
  Change from Baseline at Study Month 9 | 0.064 (0.190) | 0.015 (0.197)
  Change from Baseline at Study Month 12: number analyzed (Participants) | 79 | 32
  Change from Baseline at Study Month 12 | 0.072 (0.241) | 0.051 (0.200)
  Change from Baseline at Study Month 15: number analyzed (Participants) | 67 | 26
  Change from Baseline at Study Month 15 | 0.051 (0.209) | 0.080 (0.125)
  Change from Baseline at Study Month 18: number analyzed (Participants) | 71 | 22
  Change from Baseline at Study Month 18 | 0.094 (0.180) | 0.072 (0.188)
  Change from Baseline at Study Month 21: number analyzed (Participants) | 45 | 20
  Change from Baseline at Study Month 21 | 0.089 (0.235) | 0.110 (0.177)
  Change from Baseline at Study Month 24: number analyzed (Participants) | 33 | 12
  Change from Baseline at Study Month 24 | 0.051 (0.239) | 0.117 (0.138)
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Difference in mean change of scores from Baseline at Day 100; Test type: Superiority; p = 0.0112, Mixed Model with Repeated Measures — False Discovery Rate Methodology; Mixed Model with Repeated Measures = 0.081, 95% CI 2-sided [0.024 to 0.138]
Statistical Analysis 2: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Difference in mean change of scores from Baseline at Day 150; Test type: Superiority; p = 0.3703, Mixed Model with Repeated Measures — False Discovery Rate Methodology; Mixed Model with Repeated Measures = 0.028, 95% CI 2-sided [-0.034 to 0.091]

12. Secondary Outcome: Change From Baseline in EQ-5D-5L VAS Scale Score
Description: The EQ-5D-5L VAS is a 20-cm VAS for recording self-rated current HRQoL state and is used to describe the participants' health status on the day of the assessment. The EQ-5D-5L VAS score is recorded by each participant for his or her current HRQoL state and scored 0 ("the worst health you can imagine") to 100 ("the best health you can imagine"). The value 100 indicates improvement.
Time Frame: Baseline, Days 50, 100, 150; Months 9, 12, 15, 18, 21 and 24
Population: Participants in QoL analysis set with data available at given timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 165 | 129
Score on scale
  Score at Baseline | 72.4 (18.7) | 74.4 (20.1)
  Change from Baseline at Study Day 50: number analyzed (Participants) | 163 | 124
  Change from Baseline at Study Day 50 | -1.9 (18.7) | -4.4 (16.7)
  Change from Baseline at Study Day 100: number analyzed (Participants) | 145 | 64
  Change from Baseline at Study Day 100 | 4.0 (18.4) | -8.2 (19.8)
  Change from Baseline at Study Day 150: number analyzed (Participants) | 110 | 54
  Change from Baseline at Study Day 150 | 9.1 (19.4) | -2.2 (22.2)
  Change from Baseline at Study Month 9: number analyzed (Participants) | 88 | 39
  Change from Baseline at Study Month 9 | 11.4 (19.9) | 4.4 (19.0)
  Change from Baseline at Study Month 12: number analyzed (Participants) | 80 | 31
  Change from Baseline at Study Month 12 | 10.1 (19.9) | 6.6 (17.8)
  Change from Baseline at Study Month 15: number analyzed (Participants) | 67 | 26
  Change from Baseline at Study Month 15 | 10.7 (20.7) | 8.2 (13.7)
  Change from Baseline at Study Month 18: number analyzed (Participants) | 70 | 23
  Change from Baseline at Study Month 18 | 15.1 (17.1) | 9.3 (13.6)
  Change from Baseline at Study Month 21: number analyzed (Participants) | 45 | 20
  Change from Baseline at Study Month 21 | 14.0 (17.2) | 10.1 (14.3)
  Change from Baseline at Study Month 24: number analyzed (Participants) | 33 | 12
  Change from Baseline at Study Month 24 | 10.9 (18.8) | 12.2 (15.3)
Statistical Analysis 1: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Difference in mean change of scores from Baseline at Day 100; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures — False Discovery Rate Methodology; Mixed Model with Repeated Measures Differences in Change from Baseline; Mixed Model with Repeated Measures = 13.7, 95% CI 2-sided [8.5 to 18.8]
Statistical Analysis 2: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Difference in mean change of scores from Baseline at Day 150; Test type: Superiority; p = 0.0004, Mixed Model with Repeated Measures — False Discovery Rate Methodology; Mixed Model with Repeated Measures = 11.3, 95% CI 2-sided [5.4 to 17.1]
Statistical Analysis 3: Comparison: Axicabtagene Ciloleucel vs Standard of Care Therapy; Difference in mean change of scores from Baseline at Month 9; Test type: Superiority; p = 0.2549, Mixed Model with Repeated Measures — False Discovery Rate Methodology; Mixed Model with Repeated Measures Differences in Change from Baseline; Mixed Model with Repeated Measures = 3.8, 95% CI 2-sided [-2.3 to 10.0]

13. Secondary Outcome: Number of Participants With Post-dose Anti-Axicabtagene Ciloleucel Antibodies
Time Frame: Up to 74.9 months
Population: Participants in the Safety Analysis Set were analyzed. The Safety Analysis Set was defined as the subset of all randomized participants who received at least 1 dose of axicabtagene ciloleucel as protocol therapy or SOC chemotherapy as protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Axicabtagene Ciloleucel
Number analyzed (Participants) | 170
Participants | 0

14. Secondary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any AE that begins on or after the first dose of study treatment (axicabtagene ciloleucel infusion or SOC), excluding bridging therapy.
Time Frame: From first dose up to 61.8 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Standard of Care Therapy: Participants received 2 or 3, 21-day cycles of second-line chemotherapy regimen:
  * R-ICE: rituximab 375mg/m^2 before chemotherapy, ifosfamide 5g/m^2 24 hours infusion on Day 2 + mesna, carboplatin area under the curve (AUC) 5 Day 2, maximum dose 800mg, etoposide 100mg/m^2/day on Days 1-3;
  * R-ESHAP: rituximab 375mg/m^2 Day 1, etoposide 40mg/m^2/day IV on Days 1-4, methylprednisolone 500mg/day IV on Days 1-4 or 5, cisplatin at 25mg/m^2/day Days 1-4, cytarabine 2g/m^2 on Day 5;
  * R-GDP: rituximab 375mg/m^2 Day 1 (or Day 8), gemcitabine 1g/m^2 on Days 1 and 8, dexamethasone 40mg on Days 1-4, cisplatin 75mg/m^2 Day 1 or carboplatin AUC=5; or
  * R-DHAP: rituximab 375mg/m^2 before chemotherapy, dexamethasone 40mg/day on Days 1-4, high dose cytarabine 2g/m^2 every 12 hours for 2 doses on Day 2 following platinum, cisplatin 100mg/m^2 24 hours infusion on Day 1 or oxaliplatin 100mg/m^2.
  Participants who responded to second-line chemotherapy got high dose therapy and autologous stem cell transplant.
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 170 | 168
percentage of participants | 100.0 | 100.0

15. Secondary Outcome: Percentage of Participants With Increase in Laboratory Values Reported as Grade 3 or Higher
Description: Grading categories were determined by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Grade 1: mild, Grade 2: moderate, Grade 3: severe or medically significant, Grade 4: life-threatening. Percentages were rounded off.
Time Frame: From first dose up to 61.8 months
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 170 | 168
percentage of participants
  Hemoglobin (mmol/L) | 0 | 0
  Leukocytes (10^9/L) | 0 | 1
  Lymphocytes (10^9/L) | 0 | 0
  Alanine Aminotransferase (U/L) | 6 | 4
  Alkaline Phosphatase (U/L) | 1 | 1
  Aspartate Aminotransferase (U/L) | 6 | 2
  Bilirubin (umol/L) | 2 | 1
  Calcium (mmol/L) | 2 | 1
  Creatinine (umol/L) | 4 | 1
  Glucose (mmol/L) | 14 | 5
  Magnesium (mmol/L) | 2 | 0
  Potassium (mmol/L) | 0 | 1
  Sodium (mmol/L) | 0 | 0

16. Secondary Outcome: Percentage of Participants With Decrease in Laboratory Values Reported as Grade 3 or Higher
Description: as for outcome 15
Time Frame: From first dose up to 61.8 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel | Standard of Care Therapy
Number analyzed (Participants) | 170 | 168
percentage of participants
  Hemoglobin (mmol/L) | 41 | 44
  Leukocytes (10^9/L) | 95 | 56
  Lymphocytes (10^9/L) | 99 | 68
  Neutrophils (10^9/L) | 94 | 51
  Platelets (10^9/L) | 26 | 63
  Albumin (g/L) | 4 | 1
  Calcium (mmol/L) | 8 | 2
  Glucose (mmol/L) | 0 | 0
  Magnesium (mmol/L) | 2 | 3
  Phosphate (mmol/L) | 5 | 5
  Potassium (mmol/L) | 6 | 7
  Sodium (mmol/L) | 12 | 2

ADVERSE EVENTS:
Time Frame: All-cause mortality and Adverse events: Up to 74.9 months
Description: All-Cause Mortality: Full Analysis Set consisted of all randomized participants.
  Adverse Events: Safety Analysis Set was defined consisted of all randomized participants who received at least 1 dose of axicabtagene ciloleucel or SOC chemotherapy. Safety Retreatment Analysis Set consisted of participants retreated with axicabtagene ciloleucel.
  Data for all-cause mortality and adverse events were reported separately for initial axicabtagene ciloleucel treatment and re-treatment.
Groups:
- Axicabtagene Ciloleucel Treatment: Participants received cyclophosphamide 500 mg/m^2/day IV infusion and fludarabine 30 mg/m^2/day IV infusion conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0.
- Retreatment Axicabtagene Ciloleucel: Participants who achieved a partial response or complete response and subsequently experienced disease progression received a second course of conditioning chemotherapy (cyclophosphamide 500 mg/m^2/day IV infusion and fludarabine 30 mg/m^2/day IV infusion) for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-CD 19 CAR transduced autologous T cells/kg.
Arm/Group | Axicabtagene Ciloleucel Treatment | Standard of Care Therapy | Retreatment Axicabtagene Ciloleucel
All-Cause Mortality (participants affected / at risk) | 81/180 | 101/179 | 3/10
Serious Adverse Events (participants affected / at risk) | 96/170 | 78/168 | 2/10
Other Adverse Events (participants affected / at risk) | 170/170 | 166/168 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axicabtagene Ciloleucel Treatment (N=170) | Standard of Care Therapy (N=168) | Retreatment Axicabtagene Ciloleucel (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 22 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Heart failure with reduced ejection fraction (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0
Oesophageal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0
Incarcerated hernia (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 2 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 27 | 8 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Covid-19 (Infections and infestations) | 7 | 1 | 0
Covid-19 pneumonia (Infections and infestations) | 3 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Fungal cystitis (Infections and infestations) | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Hepatitis B reactivation (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 16 | 4 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0
Salmonella bacteraemia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 5 | 4 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 1 | 0
Wound infection (Infections and infestations) | 2 | 0 | 0
Blood stem cell harvest failure (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood fibrinogen decreased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 3 | 1
Platelet count decreased (Investigations) | 0 | 5 | 0
Troponin I increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 9 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Dyspraxia (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 17 | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 1 | 0
Hemiparesis (Nervous system disorders) | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 5 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 3 | 0
Tremor (Nervous system disorders) | 5 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 7 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 3 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 8 | 0
Faecaluria (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematopoietic stem cell mobilisation (Surgical and medical procedures) | 1 | 0 | 0
Angiopathy (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 15 | 3 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axicabtagene Ciloleucel Treatment (N=170) | Standard of Care Therapy (N=168) | Retreatment Axicabtagene Ciloleucel (N=10)
Anaemia (Blood and lymphatic system disorders) | 71 | 90 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 24 | 0
Leukopenia (Blood and lymphatic system disorders) | 9 | 6 | 0
Neutropenia (Blood and lymphatic system disorders) | 75 | 28 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 40 | 0
Sinus tachycardia (Cardiac disorders) | 58 | 16 | 4
Tachycardia (Cardiac disorders) | 13 | 10 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 11 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 11 | 0
Abdominal pain (Gastrointestinal disorders) | 22 | 23 | 1
Constipation (Gastrointestinal disorders) | 34 | 58 | 3
Diarrhoea (Gastrointestinal disorders) | 71 | 66 | 2
Dry mouth (Gastrointestinal disorders) | 16 | 8 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 14 | 0
Nausea (Gastrointestinal disorders) | 68 | 116 | 4
Stomatitis (Gastrointestinal disorders) | 4 | 29 | 0
Toothache (Gastrointestinal disorders) | 1 | 3 | 1
Vomiting (Gastrointestinal disorders) | 33 | 55 | 3
Asthenia (General disorders) | 13 | 15 | 0
Chills (General disorders) | 46 | 14 | 0
Fatigue (General disorders) | 69 | 87 | 2
Malaise (General disorders) | 15 | 9 | 1
Mucosal inflammation (General disorders) | 1 | 15 | 0
Oedema peripheral (General disorders) | 20 | 28 | 0
Pain (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 149 | 40 | 9
Hypertransaminasaemia (Hepatobiliary disorders) | 11 | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 19 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 14 | 5 | 0
Pneumonia (Infections and infestations) | 2 | 5 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 5 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 12 | 0
Alanine aminotransferase increased (Investigations) | 31 | 16 | 2
Aspartate aminotransferase increased (Investigations) | 24 | 15 | 1
Blood alkaline phosphatase increased (Investigations) | 10 | 14 | 0
Blood bilirubin increased (Investigations) | 5 | 2 | 1
Blood creatinine increased (Investigations) | 10 | 15 | 0
C-reactive protein increased (Investigations) | 15 | 4 | 0
Lymphocyte count decreased (Investigations) | 31 | 21 | 3
Neutrophil count decreased (Investigations) | 51 | 45 | 5
Platelet count decreased (Investigations) | 30 | 64 | 1
Serum ferritin increased (Investigations) | 15 | 0 | 0
Weight decreased (Investigations) | 11 | 6 | 1
Weight increased (Investigations) | 1 | 12 | 0
White blood cell count decreased (Investigations) | 46 | 37 | 4
Decreased appetite (Metabolism and nutrition disorders) | 42 | 41 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 7 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 27 | 17 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 22 | 12 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 27 | 17 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 44 | 47 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 | 34 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 19 | 7 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 45 | 29 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 14 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 23 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 14 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 18 | 11 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 7 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 9 | 0
Aphasia (Nervous system disorders) | 31 | 0 | 1
Dizziness (Nervous system disorders) | 36 | 21 | 0
Dysgeusia (Nervous system disorders) | 4 | 14 | 0
Encephalopathy (Nervous system disorders) | 18 | 1 | 0
Headache (Nervous system disorders) | 69 | 43 | 6
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 7 | 14 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 10 | 0
Somnolence (Nervous system disorders) | 14 | 2 | 0
Tremor (Nervous system disorders) | 41 | 1 | 1
Anxiety (Psychiatric disorders) | 11 | 14 | 2
Confusional state (Psychiatric disorders) | 34 | 4 | 0
Insomnia (Psychiatric disorders) | 21 | 26 | 0
Acute kidney injury (Renal and urinary disorders) | 12 | 16 | 0
Micturition urgency (Renal and urinary disorders) | 4 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 12 | 5 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 18 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 20 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 21 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 34 | 13 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 14 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 10 | 0
Erythema (Skin and subcutaneous tissue disorders) | 10 | 3 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 9 | 1
Embolism (Vascular disorders) | 1 | 1 | 1
Hypertension (Vascular disorders) | 15 | 15 | 0
Hypotension (Vascular disorders) | 66 | 23 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT03391466/Prot_002.pdf
  • Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT03391466/SAP_001.pdf